CLINICAL TRIAL: NCT06648486
Title: Evaluation of a Portable Isokinetic Knee Training Device for Quadriceps Rehabilitation in Children With SMA
Brief Title: Robot-assisted Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beihang University (Other)
Responsible Party: Principal Investigator, Yuan Fuzhen, Principle Investigator, Peking University Third Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-973-02
Record Dates: First submitted 2024-10-03; First posted 2024-10-18 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Spinal Muscular Atrophy (SMA)
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Masking Description: 7 Children with SMA, 6 Healthy Children as comparison
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Robot-assisted Rehabilitation for children with SMA type II (Experimental)
  Interventions: Device: With the assistance of wearable isokinetic training robot （ 7 children with SMA type II）
- Non-robot-assisted Rehabilitation for children with SMA type II (No Intervention): Prior to the intervention, all participants will complete a 1.5-month "Stage 0" observation period with no robot assistance. During this time, we will record each child's sit-to-stand angle to establish baseline (control) measurements.
- Biomechanical measures for healthy children (No Intervention): A single set of biomechanical measurements will be taken from healthy children to serve as a reference baseline.

INTERVENTIONS:
Device: With the assistance of wearable isokinetic training robot （ 7 children with SMA type II） — A child with SMA will use a wearable isokinetic training robot to train the knee joint for three stages. ( Stage 1: 1.5 months=30 sessions; Stage 2 (follow up): 1.5 months=18 sessions, Stage 3(follow up) = 0 session)
  Arms: Robot-assisted Rehabilitation for children with SMA type II

SUMMARY:
The goal of this clinical trial is to evaluate the long-term effects of isokinetic rehabilitation training in patients with spinal muscular atrophy (SMA). The main question it aims to answer is:

• Does isokinetic training at fixed angular velocity improve muscle strength and functional recovery in SMA patients?

Participants will:

* Perform isokinetic training using a portable device with a fixed angular velocity.
* Undergo long-term rehabilitation sessions, with assessments of muscle strength and overall functional improvement over the training period.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 6-12 years old.
2. Diagnosed with Type II Spinal Muscular Atrophy (SMA).

Exclusion Criteria:

1. Participants with severe comorbidities, implanted medical devices preventing MRI or claustrophobia were excluded from the study.
2. Refusal to provide informed consent or inability to complete the entire study protocol, among other factors;
3. Uncontrolled hypertension (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥95 mmHg) or congestive heart failure classified as New York Heart Association (NYHA) Class III or IV;
4. Cognitively impaired or unable to comprehend the requirements of study participation.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in cross sectional area of quadriceps | Baseline, after 1.5 months, after 3 months and after 4 months
  Using Magnetic Resonance Imaging (MRI)
Change in longitudinal cross-sectional width of quadriceps | Baseline, after 1.5 months, after 3 months and after 4 months
  Using Magnetic Resonance Imaging (MRI)
Change in peak torque | Baseline, after 1.5 months, after 3 months and after 4 months
  Using isokinetic training robot to measure.
Change in average torque | Baseline, after 1.5 months, after 3 months and after 4 months
  Using isokinetic training robot to measure.
Change in work of knee | Baseline, after 1.5 months, after 3 months and after 4 months
  Work = Torque * Speed
Change in Surface Electromyography (sEMG) | Baseline, after 1.5 months, after 3 months and after 4 months
Change in Nerve conduction | Baseline, after 1.5 months, after 3 months and after 4 months
  Nerve Conduction Velocity Testing System

SECONDARY OUTCOMES:
Change in weight | Baseline, after 1.5 months, after 3 months and after 4 months
Change in height | Baseline, after 1.5 months, after 3 months and after 4 months
Change in joint angle | Baseline, after 1.5 months, after 3 months and after 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-12-13): https://cdn.clinicaltrials.gov/large-docs/86/NCT06648486/Prot_SAP_ICF_002.pdf